CLINICAL TRIAL: NCT03075670
Title: A Trial Comparing the Pharmacokinetics of Nonacog Beta Pegol (N9-GP) and ALPROLIX® in Patients With Haemophilia B
Brief Title: A Trial Comparing Nonacog Beta Pegol (N9-GP) and ALPROLIX® in Patients With Haemophilia B
Acronym: paradigm™7
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NN7999-4260; 2016-001149-25 (EudraCT Number); U1111-1180-7154 (Other: World Health Organization (WHO))
Record Dates: First submitted 2017-03-03; First posted 2017-03-09 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Congenital Bleeding Disorder; Haemophilia B
MeSH Terms: conditions — Hemophilia B | interventions — factor IX Fc fusion protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- N9-GP (Experimental)
  Interventions: Drug: N9-GP
- ALPROLIX® (Active Comparator)
  Interventions: Drug: ALPROLIX®

INTERVENTIONS:
Drug: N9-GP — A single dose of 50 IU/kg for intravenous (i.v.) injection
  Arms: N9-GP
Drug: ALPROLIX® — A single dose of 50 IU/kg for intravenous (i.v.) injection
  Arms: ALPROLIX®

SUMMARY:
This trial is conducted in Europe and the United States of America. The aim of this trial is to compare the pharmacokinetics (the exposure of the trial drug in the body) of nonacog beta pegol (N9-GP) and ALPROLIX® in patients with haemophilia B.

ELIGIBILITY:
Inclusion Criteria:

* Male, aged 18-70 years (both inclusive) at the time of signing informed consent
* Patients with the diagnosis of congenital haemophilia B with factor IX activity below or equal to 2%, based on medical records
* History of more than 150 exposures days to any factor IX containing products

Exclusion Criteria:

* Known history of factor IX inhibitors
* Inhibitors to factor IX (above or equal to 0.6 BU) at screening measured by the Nijmegen modified Bethesda method
* Immunocompromised (CD4+ T cells below or equal to 200/μL)
* Known congenital or acquired coagulation disorders other than haemophilia B
* Body mass index above 35 kg/m^²

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-03-07 (Actual); Primary Completion 2017-12-08 (Actual); Study Completion 2017-12-08 (Actual)

PRIMARY OUTCOMES:
Area under the factor IX activity-time curve from 0 to infinity dose-normalised to 50 IU/kg | From time 0 (dosing) up to 240 hours post-dose
  Calculated based on plasma FIX activity measured in blood

SECONDARY OUTCOMES:
Maximum activity dose-normalised to 50 IU/kg (Cmax,norm) | From time 0 (dosing) up to 240 hours post-dose
  Calculated based on plasma FIX activity measured in blood
Incremental recovery at 30 minutes (IR30min) | At 30 minutes
  Calculated based on plasma FIX activity measured in blood
Terminal half-life (t½) | From time 0 (dosing) up to 240 hours post-dose
  Calculated based on plasma FIX activity measured in blood
Clearance (CL) | From time 0 (dosing) up to 240 hours post-dose
  Calculated based on plasma FIX activity measured in blood
Area under the activity-time curve | From time 0 (dosing) up to 240 hours post-dose
  Calculated based on plasma FIX activity measured in blood
Maximum activity (Cmax) | From time 0 (dosing) up to 240 hours post-dose
  Calculated based on plasma FIX activity measured in blood
Activity at 30 minutes (C30min) | at 30 minutes
  Calculated based on plasma FIX activity measured in blood
Activity at 168 hours (C168h) | At 168 hours
  Calculated based on plasma FIX activity measured in blood
Incremental recovery at maximum activity (IRCmax) | From time 0 (dosing) up to 240 hours post-dose
  Calculated based on plasma FIX activity measured in blood
Time of maximum activity (tmax) | From time 0 (dosing) up to 240 hours post-dose
  Calculated based on plasma FIX activity measured in blood
Apparent volume of distribution during terminal phase (Vz) | From time 0 (dosing) up to 240 hours post-dose
  Calculated based on plasma FIX activity measured in blood
Apparent volume of distribution at steady-state (Vss) | From time 0 (dosing) up to 240 hours post-dose
  Calculated based on plasma FIX activity measured in blood
Mean residence time (MRT) | From time 0 (dosing) up to 240 hours post-dose
  Calculated based on plasma FIX activity measured in blood
Terminal elimination rate constant | From time 0 (dosing) up to 240 hours post-dose
  Calculated based on plasma FIX activity measured in blood
Area under the activity-time curve from 0 to infinity | From time 0 (dosing) up to 240 hours post-dose
  Calculated based on plasma FIX activity measured in blood
Area under the activity-time curve from 0 to t last | From time 0 (dosing) up to 240 hours post-dose
  Calculated based on plasma FIX activity measured in blood
Number of adverse events | From time 0 (dosing) up to 240 hours post-dose
  Count and % of Adverse events

CONTACTS AND LOCATIONS:
Locations (12):
- United States (7):
  - Novo Nordisk Investigational Site, Phoenix, Arizona
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Peoria, Illinois
  - Novo Nordisk Investigational Site, East Lansing, Michigan
  - Novo Nordisk Investigational Site, Rochester, Minnesota
  - Novo Nordisk Investigational Site, Oklahoma City, Oklahoma
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
- Germany (4):
  - Novo Nordisk Investigational Site, Berlin
  - Novo Nordisk Investigational Site, Duisburg
  - Novo Nordisk Investigational Site, Hanover
  - Novo Nordisk Investigational Site, Mörfelden-Walldorf
- Novo Nordisk Investigational Site, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com

REFERENCES:
- [Derived] Escuriola Ettingshausen C, Hegemann I, Simpson ML, Cuker A, Kulkarni R, Pruthi RK, Garly ML, Meldgaard RM, Persson P, Klamroth R. Favorable pharmacokinetics in hemophilia B for nonacog beta pegol versus recombinant factor IX-Fc fusion protein: A randomized trial. Res Pract Thromb Haemost. 2019 Mar 23;3(2):268-276. doi: 10.1002/rth2.12192. eCollection 2019 Apr. PMID 31011711